CLINICAL TRIAL: NCT07291375
Title: The Effect of Low Dose Oral Amlodipine in Renal Protection From Contrast Induced Nephropathy in Diabetic Patients in Intensive Care Unit
Brief Title: Role of Amlodipine in Reduction of CIN
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Andrew Samy Shafeek Shehata, Andrew Samy Shafeek, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Amlodipine role in CIN
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Contrast-induced Nephropathy
MeSH Terms: interventions — Calcium Channel Blockers; Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): this group who undergoing iv contrast will receive hydration only
  Interventions: Other: Hydration
- Amlodipine group (Other): this group will receive hydration and amlodipine
  Interventions: Drug: Calcium channel blocker; Other: Hydration

INTERVENTIONS:
Drug: Calcium channel blocker — amlodipine group will receive low dose oral amlodipine ( 5 mg ) before iv contrast and every 12 hour for 48 hour
  Other Names: amlodipine ( 5mg)
  Arms: Amlodipine group
Other: Hydration — before the procedure patients will recieve iv bolus of 250 ml saline followed by continous infusion of 100 ml/h of normal saline

SUMMARY:
The aim is to assess the benefit of low dose oral amlodipine in renal protection from contrast induced nephropathy in diabetic patients in intensive care unit

ELIGIBILITY:
Inclusion Criteria:

* adult patients of both sexes (18:70) diabetic patients with serum creatinine below 1.2 hemodynamically stable patients ASA physical status 2,3

Exclusion Criteria:

* patient refusal patients of chronic kidney diseases NPO patients serum creatinine above 1.2 Hypertensive patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
measuring serum creatinine level | baseline
  measuring serum creatinine level before the procedure and every day for 48 hours after